CLINICAL TRIAL: NCT07167316
Title: Phase I, Randomized, Placebo-Controlled Study on the Role of the LC-NA System in Experimental Sleep Fragmentation With Buccal Dexmedetomidine.
Brief Title: The Role of the LC-NA System in Experimental Sleep Fragmentation
Acronym: DMTN_FragSleep
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hans-Peter Landolt (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor-Investigator, Hans-Peter Landolt, Prof. Dr. sc. nat., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2025-01005
Record Dates: First submitted 2025-07-17; First posted 2025-09-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-09

CONDITIONS: The Role of the LC-NA System in Sleep Regulation
Keywords: Cross-Over; placebo controlled; randomized; sleep disturbance; auditory stimulation; healthy; Stress; LC-NA; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Parasomnias | interventions — Acoustic Stimulation

STUDY DESIGN:
Intervention Model Description: Each participant will first spend a screening night to adapt to the sleep laboratory environment, followed by a baseline night without any interventions. Subsequently, they will complete three experimental nights, during which sleep will be disrupted using auditory stimulation. On each of these nights, participants will receive either a high dose, a low dose of dexmedetomidine, or a placebo. The order in which these three conditions are administered will be randomized across participants. In a second part of the study, participants will spend three nights again receiving the high dose, low dose, or placebo in randomized order. During these nights, blood samples will be collected for pharmacokinetic analyses, and additional physiological measures will be recorded to assess pharmacodynamic effects.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Low Dose (Experimental): Experimental: 64 µg Dexmedetomidine
  Interventions: Drug: DMTN
- High Dose (Experimental): Experimental: 96 µg Dexmedetomidine
  Interventions: Drug: DMTN
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placbo
- Low Dose + Auditory Stimulation (Experimental): Experimental: 64 µg Dexmedetomidine + Auditory Stimulation
  Interventions: Drug: DMTN; Other: Auditory Stimulation
- High Dose + Auditory Stimulation (Experimental): Experimental: 96 µg Dexmedetomidine + Auditory Stimulation
  Interventions: Drug: DMTN; Other: Auditory Stimulation
- Placebo + Auditory Stimulation (Placebo Comparator): Placebo + Auditory Stimulation
  Interventions: Other: Auditory Stimulation; Drug: Placbo

INTERVENTIONS:
Drug: DMTN — Dexmedetomidine is a highly selective alpha-2 adrenergic receptor agonist that reduces the release of norepinephrine by inhibiting activity in the locus coeruleus, a key brain region involved in arousal and stress responses. In this study, dexmedetomidine will be administered as an oro-dispersible tablet applied buccally, allowing for rapid absorption through the oral mucosa.
  Arms: High Dose; High Dose + Auditory Stimulation; Low Dose; Low Dose + Auditory Stimulation
Other: Auditory Stimulation — Auditory tones will be presented throughout the night at individually calibrated intensities, adjusted to each participant's hearing threshold, in order to induce controlled sleep fragmentation without full awakenings.
  Arms: High Dose + Auditory Stimulation; Low Dose + Auditory Stimulation; Placebo + Auditory Stimulation
Drug: Placbo — Oro-dispersible placebo tablet identical in appearance and packaging to the active Dexmedetomidine tablet.
  Arms: Placebo; Placebo + Auditory Stimulation

SUMMARY:
Sleep-wake regulation affects every person's life, yet the molecular mechanisms underlying these processes remain poorly understood. In particular, the microstructure of sleep has not been sufficiently studied to explain how sleep produces a feeling of restoration the following morning. Stress also plays a significant role in sleep regulation. This study aims to investigate the role of norepinephrine in these processes.

DETAILED DESCRIPTION:
Following a screening night and a baseline sleep recording, participants undergo three experimental nights in the sleep laboratory. On each of these nights, sleep is intentionally disrupted using auditory stimuli to induce fragmentation. To investigate potential counteracting effects on sleep quality, participants receive either a low dose (64 µg), a high dose (96 µg) of dexmedetomidine (DMTN)-a compound known to reduce norepinephrine levels-or a placebo. All participants experience each condition in a randomized, double-blind, crossover design, with the sequence of administration varying between individuals. Neither the participants nor the study team are aware of the assigned condition on any given night.

In a second part of the study, three additional nights are conducted to assess the pharmacokinetics and pharmacodynamics of dexmedetomidine. During these nights, participants again receive either the low dose (64 µg), high dose (96 µg), or placebo (in randomized order). Blood samples are collected at multiple time points to characterize the compound's pharmacokinetic profile, and additional physiological outcomes are measured to evaluate pharmacodynamic effects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 35 years (inclusive)
* Body-Mass-Index (BMI): 18.5 < BMI < 25
* Non-nicotine user status
* Habitual consumption of 5 or fewer alcoholic beverages / week
* Habitual consumption of 3 or fewer caffeinated beverages / day
* Habitual average sleep duration 7-9 h / night
* Normal or corrected-to-normal vision
* Insomnia severity Index (ISI) Score: ISI < 8
* Ability to understand and speak German language
* Normal hearing ability (applies only to Sleep Study Part)
* Ability and willingness to provide informed consent as documented by dated signature

Exclusion Criteria:

* Present use of medication that may interfere with sleep or study drugs
* Travel across 3 or more time zones within 3 months of study start
* Habitual napping
* Extreme chronotype, determined by reduced Morningness-Eveningness Questionnaire (rMEQ) score: 8 < rMEQ > 21)
* Shift working within 2 weeks prior to the screening visit
* History of or presence of a trauma- or stressor-related disorder
* Serious acute or chronic neurological, mental, or general medical conditions that, in the opinion of the investigator, may pose a risk to participation or affect study measurements
* History of or presence of a sleep wake disorder
* Use of illicit drugs (positive urinary drug screening)
* Male participants who are not vasectomised for at least 6 months prior to dosing and who are sexually active with a female partner of childbearing potential not willing to use one of the following acceptable contraceptive methods from the first dose and for 3 months after the last dose:

Use of condom and/or hormonal contraceptive (e.g., oral, patch, depot injection, implant, vaginal ring, intrauterine device) or non-hormonal intrauterine device used for at least 4 weeks prior to sexual intercourse for the female partner;

* Male participants (including men who have had a vasectomy) with a pregnant partner not willing to use a condom from the first dose and for 3 months after the last dose.
* Male participants not willing to abstain from sperm donation for 3 months after the last dose
* Females of childbearing potential who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomised at least 6 months prior to the first study drug administration) not willing to use one of the following acceptable contraceptive methods throughout the study and for at least 3 months after the last study drug administration:

Simultaneous use of condom and hormonal contraceptive (e.g., oral, patch, depot injection, implant, vaginal ring, intrauterine device) or non-hormonal intrauterine device used for at least 4 weeks prior to sexual intercourse for the female partner;

- Females of non-childbearing potential who are neither: Post-menopausal (status defined as an absence of menses for at least 12 months prior to the first study drug administration); or Surgically sterilized (complete hysterectomy or bilateral oophorectomy at least 3 months prior to the first study drug administration)

* Faints at the sight of blood (applies only for the pharmacokinetic-part of the study)
* Has participated in a study < 30 days or a study such as this (i.e., experimental trauma) at all.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Total Sleep Time (TST) | Baseline Night, Experimental Night 1, Experimental Night 2, Experimental Night 3
  The total amount of time spent in all sleep stages (N1, N2, N3, and REM) combined, measured in minutes.
Change in Wake After Sleep Onset (WASO) | Baseline Night, Experimental Night 1, Experimental Night 2, Experimental Night 3
  The total time spent awake in minutes after sleep has been initiated and before the final awakening.
Change in Sleep Efficiency | Baseline Night, Experimental Night 1, Experimental Night 2, Experimental Night 3
  The percentage of time spent asleep relative to the total time spent in bed (Total Sleep Time / Time in Bed * 100).
Change in Sleep Onset Latency (SOL) | Baseline Night, Experimental Night 1, Experimental Night 2, Experimental Night 3
  The time in minutes from "lights out" to the first epoch of any sleep stage.
Percentage of Time in N1, N2, N3 and REM-Sleep | Baseline Night, Experimental Night 1, Experimental Night 2, Experimental Night 3
  The proportion of Total Sleep Time spent in Stage N1, N2, N3 and REM-Sleep.
Change in Arousal Index | Baseline Night, Experimental Night 1, Experimental Night 2, Experimental Night 3
  The number of EEG arousals per hour of sleep.
Maximum Plasma Concentration (Cmax) of Dexmedetomidine | Up to 24 hours post-dose on Experimental Night 1, Experimental Night 2, and Experimental Night 3
  The maximum observed concentration of dexmedetomidine in plasma following administration, determined from serial blood sampling.
Time to Maximum Plasma Concentration (Tmax) of Dexmedetomidine | Up to 24 hours post-dose on Experimental Night 1, Experimental Night 2, and Experimental Night 3
  The time at which the maximum plasma concentration (Cmax) of dexmedetomidine is observed following administration.
Area Under the Plasma Concentration-Time Curve From Time 0 to Last Measurable Point (AUC0-t) of Dexmedetomidine | Up to 24 hours post-dose on Experimental Night 1, Experimental Night 2, and Experimental Night 3
  The cumulative drug exposure over time, calculated as the area under the dexmedetomidine plasma concentration versus time curve from the time of dosing to the last quantifiable plasma concentration.
Change in Plasma Noradrenaline Concentration | Up to 24 hours post-dose on Experimental Night 1, Experimental Night 2, and Experimental Night 3
  Assessment of the change in endogenous noradrenaline levels in plasma, measured from samples collected at predetermined timepoints following intervention.

SECONDARY OUTCOMES:
Dim Light Melatonin Onset (DLMO) | Evening after Experimental Night 1, Evening after Experimental Night 2, Evening after Experimental Night 3
  The clock time at which the concentration of salivary melatonin first exceeds a calculated threshold, determined by serial sampling in dim light conditions. DLMO is a key marker of circadian phase.
Change in Autonomic Arousal Measured by Pupillometry | Pre-dose, 15 minutes post-dose, 2 hours post-dose (only PK-Part), 4 hours post-dose (only PK-Part), 15 minutes after lights on.
  To quantify autonomic arousal, pupillometry will be performed at different schedules. During sleep-focused visits, assessments are at pre-dose, 15 minutes post-dose, and 15 minutes after lights on. During pharmacokinetic-focused visits, additional assessments are made at 2 and 4 hours post-dose. Autonomic arousal will be reported as a single index derived from pupil diameter and its fluctuations.
Change in Heart Rate Variable | Baseline Night, Experimental Night 1, Experimental Night 2, Experimental Night 3
  Heart rate variables, will be continuously monitored to assess autonomic nervous system regulation.
Resting-state EEG spectral analysis | Pre-sleep (evening) and post-sleep (morning) at the baseline night and each of the 3 overnight experimental visits (together with the "Change in Autonomic Arousal Measured by Pupillometry" acquisition).
  Wake-state EEG will be recorded before and after sleep to assess changes in power spectral density, especially in alpha and theta bands.
Nocturnal thermoregulation | Baseline Night, Experimental Night 1, Experimental Night 2, Experimental Night 3
  Body temperature will be continuously monitored to evaluate effects of Dexmedetomidine on thermoregulation.
Pre-sleep arousal levels (PSAS) | Morning of Baseline Night, Morning of Experimental Night 1, Morning of Experimental Night 2, Morning of Experimental Night 3
  The Pre-Sleep Arousal Scale (PSAS, score range 16 - 80, with higher scores indicating higher levels of arousal) will be administered to assess cognitive and somatic arousal prior to bedtime.
Sedation depth (OAAS scale) | Completed at each of the 3 overnight experimental visits similar to the blood sampling timepoints in the sleep opportunity window.
  Observer-rated sedation will be assessed using the Observer's Assessment of Alertness/Sedation Scale (score 1 - 5).
Mood states (POMS-16 and A-SIQ) | Morning following Baseline Night, Morning following Experimental Night 1, Morning following Experimental Night 2, Morning following Experimental Night 3
  Mood and sleep inertia will be evaluated using the 16-item Profile of Mood States (POMS-16, 16 items from 0-4; assesses mood across five subscales, with higher scores indicating greater intensity except for vigor) and the Acute Sleep Inertia Questionnaire (A-SIQ, 22 items from -3 - +3, with higher scores indicate more sleep inertia and 1 item with visual analoge scale) upon awakening.
State-Trait Anxiety Inventory (STAI) | Morning following Baseline Night, Morning following Experimental Night 1, Morning following Experimental Night 2, Morning following Experimental Night 3
  Trait and state anxiety will be assessed via the STAI-Y1 (STAI-Y1, 20 items from 1-4; higher scores reflect greater momentary anxiety) questionnaire to explore mood modulation effects of the experimental sleep fragmentation and Dexmedetomidine.
Psychomotor vigilance (PVT) | Morning following Baseline Night, Morning following Experimental Night 1, Morning following Experimental Night 2, Morning following Experimental Night 3
  Vigilance performance will be assessed using the Psychomotor Vigilance Task (PVT) upon awakening.
Number of Participants with Orthostatic Intolerance as Defined by Schellong Test Criteria | Morning following Baseline Night, Morning following Experimental Night 1, Morning following Experimental Night 2, Morning following Experimental Night 3
  The number of participants who are unable to complete the full duration of the Schellong test or exhibit clear signs of intolerance. This is defined as the occurrence of any of the following: participant-reported dizziness or pre-syncope requiring termination of the test; investigator-observed excessive swaying or stumbling requiring intervention; or early termination of the test at the participant's request.
Number of Participants Exhibiting Clinically Significant Gait Instability During a Standardized Gait Task | In the morning after 8 hours sleep opportunity window of the baseline night and each of the 3 overnight experimental visits. For the PK part additional timepoints (2 & 4 hours post dosing) will be measured during sleep opportunity window of 8 hours.
  Postural stability and adaptation during walking will be assessed via a standardized gait task. Clinically significant instability is defined as the occurrence of any of the following during the task: any stumble, trip, or loss of balance; requiring physical assistance or support from an external surface (e.g., a wall); or an inability to complete the prescribed walking task as instructed.
Change in Power of EEG Infra-Slow Oscillations (<0.1 Hz) During NREM Sleep | Baseline Night, Experimental Night 1, Experimental Night 2, Experimental Night 3
  The power spectral density of EEG activity (measured in μV²/Hz) in the infra-slow frequency band (<0.1 Hz), calculated from overnight polysomnography (PSG) recordings during NREM sleep. The change from the placebo condition to the DMTN condition will be calculated to assess the drug's effect on rhythmic noradrenergic signalling.
Change in Blood Oxygen Saturation (SpO2) | Continuously during each 3 of the the pharmacokinetic overnight experimental visits.
  Peripheral blood oxygen saturation (SpO2), measured as a percentage, will be continuously monitored via pulse oximetry during the pharmacokinetic (PK) study visits.
Change in Systolic Blood Pressure | Evening and Morning of Baseline Night, Evening and Morning of Experimental Night 1, Evening and Morning of Experimental Night 2, Evening and Morning of Experimental Night 3
  Systolic blood pressure (SBP), measured in mmHg, will be assessed at discrete time points in the evening and morning to evaluate autonomic changes.
Change in Diastolic Blood Pressure | Evening and Morning of Baseline Night, Evening and Morning of Experimental Night 1, Evening and Morning of Experimental Night 2, Evening and Morning of Experimental Night 3
  Diastolic blood pressure (DBP), measured in mmHg, will be assessed at discrete time points in the evening and morning to evaluate autonomic changes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Institute of Pharmacology and Toxicology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Any disclosure of information to individuals not directly involved in the study must be approved by the owner of the data.

REFERENCES:
- See also: Paper of our previous research project, providing the background for the current study — https://pmc.ncbi.nlm.nih.gov/articles/PMC11801451/